CLINICAL TRIAL: NCT06379620
Title: Pilot Open Label Use of the Hi-OXSR to Increase PaCO2 for the Treatment of Post COVID-19 Cognitive Dysfunction
Brief Title: Pilot Open Label Use of the Hi-OXSR for the Treatment of Post COVID-19 Cognitive Dysfunction
Acronym: Hi-OXSR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-5544
Record Dates: First submitted 2024-04-22; First posted 2024-04-23 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Post COVID-19 Condition
Keywords: cognitive dysfunction; post-COVID condition; long COVID; SARS-CoV2
MeSH Terms: conditions — Cognitive Dysfunction; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: This is an open label, pilot treatment study. Screening data will be reviewed to determine subject eligibility. Upon successful completion of all screening procedures, subject will be considered eligible for enrollment.
  The subject will self-administer oxygen gas at 1to 3LPM via a Hi-OxSR Sequential Rebreathing mask, twice a day for 30 minutes with ventilation supplemented by the subject's rebreathed exhaled air. Total treatment is for 14 days. Subjects will be asked to return to the clinic for additional evaluations on Days 15 and 45.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Hi-OXSR group (Experimental): Oxygen gas at 1 to 3LPM via a Hi-OxSR Sequential Rebreathing mask (oxygen concentrator), twice a day for 30 minutes with increased inspired CO2 concentration produced by having the subject rebreathe some of their exhaled air. Total treatment is for 14 days.
  Interventions: Device: Hi-OxSR Sequential Rebreathing mask (oxygen concentrator)

INTERVENTIONS:
Device: Hi-OxSR Sequential Rebreathing mask (oxygen concentrator) — Subjects will self-administer oxygen gas at 1to 3LPM via a Hi-OxSR Sequential Rebreathing mask (oxygen concentrator), twice a day for 30 minutes with ventilation supplemented by the subject's rebreathed exhaled air. Total treatment is for 14 days

SUMMARY:
During the worldwide COVID-19 pandemic a large number patients reported different functional complaints one month or later after recovery from the acute infection. This entity had a number of names including "long-COVID" or "post COVID condition". Long-COVID is on the rise and no effective treatment exists yet to improve cognitive function. Recent research has shown that people with even mild COVID had a greater decline in executive function, notably in their ability to perform complex tasks. What drives post-COVID cognitive changes is still a mystery and there are no effective treatments available. One hypothesis is that there is persistent immune activation resulting in reduction in cerebral blood flow. There is evidence that increased CO2 may decrease inflammation, and decreased CO2 may increase inflammation.

Objectives: The primary objective of this pilot study is to assess the safety and tolerability of the use of Hi-OX sequential rebreathing for the treatment of post-COVID cognitive dysfunction. The secondary objective is to identify the effects of the use of the Hi-OX rebreathing treatment in changing post-COVID cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent.
2. Previously diagnosed with cognitive dysfunction following recovery from COVID.
3. Not pregnant at time of study.
4. Oxygen saturation on room air ≥92% at screening.
5. Willing and able to comply with the treatment schedule and procedures.

Exclusion Criteria:

1. History of cognitive dysfunction prior to COVID infection
2. Hospitalization for the treatment of COVID
3. Participating in another investigational trial or the use of an investigational drug within 30 days of screening
4. For individuals of childbearing potential:

   positive pregnancy test at screening or lactating or unwilling to practice a medically acceptable form of contraception from screening to Day 14 (acceptable forms of contraception: abstinence, hormonal birth control, intrauterine device, or barrier method plus a spermicidal agent)
5. History of pulmonary hypertension
6. History of narcolepsy
7. Moderate to severe COPD
8. Interstitial Pulmonary Fibrosis
9. End-tidal PCO2 >55 mmHg during training treatment
10. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Safety of use of Hi-OX sequential rebreathing device | 45 days
  Any unanticipated adverse events reporting

CONTACTS AND LOCATIONS:
Overall Officials: Angela Cheung, Md, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada